CLINICAL TRIAL: NCT05658627
Title: Effect of Hamstring Active Release Technique in Cervicogenic Headache
Brief Title: Hamstring Active Release Technique in Cervicogenic Headache
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samar Ahmed El Sayed Mohammed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003916
Record Dates: First submitted 2022-12-12; First posted 2022-12-21 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Cervicogenic Headache
Keywords: active release technique and cervicogenic headache
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1- control group (Active Comparator): conventional physical therapy (ultrasound therapy- stretching exercise- strengthening exercise)
  Interventions: Other: conventional therapy
- 2- Experimental group (Experimental): Active release technique for hamstring+ conventional physical therapy(ultrasound therapy- stretching exercise- strengthening exercise)
  Interventions: Other: active release technique; Other: conventional therapy

INTERVENTIONS:
Other: active release technique — Hamstring active release technique-
  Arms: 2- Experimental group
Other: conventional therapy — ultrasound therapy - stretching Exercise - Strengthening Exercise -

SUMMARY:
It has been suggested that the suboccipital muscles are a causative factor in both cervicogenic neck pain and headache. Hamstrings and sub-occipital muscles are connected by a neural system and sub-occipital muscles pass through the dura Mater. Increased tension and shortening of the hamstring's muscles can cause neck and shoulder pain. In addition, when the muscles around the neck are tensed, the muscles in the limbs are also tensed, so that if the tone of the hamstring muscles is decreased, SLR test score increased, and the tone of the sub-occipital muscles is reduced. Active release technique is found to have an effect on hamstring flexibility.

DETAILED DESCRIPTION:
Cervicogenic Headache (CGH) is a secondary and often unilateral headache that is known by referring pain from soft or hard cervical structures to occipital, temporal and frontal regions. There are some fascial connections between suboccipital muscles with dura mater and C2 vertebra. Presumably, fascial restriction in one part of the body causes unusual stress in other parts of the body due to fascial continuity. It has demonstrated that increased tension and shortening of the hamstring's muscles can cause neck and shoulder pain. This occurs because the superficial fascial back line of the myofascial chain connects from the neck to the lower extremity, and the soft tissue in the cervical spine links the dura and suboccipital muscle fascia. Therefore, it is probable that if the tone of the hamstring muscles is decreased (passively, with a fascial treatment or with active movements), the tone of the knee flexors (hamstring muscles) is reduced and the amplitude of hip flexion is increased, thereby increasing the straight leg raise (SLR) test score. Active release technique (ART) is a type of manual therapy used for treating soft tissue injuries. Problems with muscles, tendons, ligaments, fascia and nerves are successfully treated with it and is found to have an effect on hamstring flexibility.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral headache (in the same side) related by pain, movement and sustaining position of neck started from the occiput spread to the tempro-frontal region for more than 3 months.
* Pain and tenderness at the upper cervical segment's palpation.
* Movement restriction in cervical region, especially in the upper cervical rotation.
* Positive SLR test for hamstring muscle less than 80◦.

Exclusion Criteria:

* Malignancy.
* Other types of headaches, including migraine, tension type, other serious headaches.
* History of head and neck trauma or surgery.
* Pregnancy.
* Physiotherapy for headache in the last 3 months.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Assess the change in pain intensity level | Before treatment and after 4 weeks treatment
  The visual analogue scale (VAS) is a widely utilized pain intensity level assessment instrument in rehabilitation.VAS is typically composed of a 100 mm horizontal line attached with two opposed labels, the left end marked "no pain" and the right end "severe intolerable pain".Patients will mark a score on the scale by a vertical line.
Assess the change in headache severity | Before treatment and after 4 weeks treatment
  The headache impact test (HIT-6) : is a tool that subjectively evaluates the frequency of a patient's headache. The lowest score is 36, and the highest score is 78 for six items.Usually, if the score is over 59, it means the patient's daily life is severely affected by the headache.
Assess the change in pressure pain threshold | Before treatment and after 4 weeks treatment
  Pressure algometry will be used to evaluate the (PPT) for suboccipital and hamstring muscles.In the prone position, the physician will apply 1 kg/s of pressure directly to suboccipital and hamstring muscles, the participant will speak up at the point where the pressure evoke a painful sensation, and the instantaneous value will be recorded as the PPT.

SECONDARY OUTCOMES:
Assess the change in Cervical flexion rotation test | Before treatment and after 4 weeks treatment
  By the cervical range of motion (CROM) instrument placed on the head.The evaluator will perform maximum flexion of the cervical spine followed by a rotation to each side.Each measurement will be repeated 3 times at 30 s intervals. The mean value obtained from the 3 trials will be used for data analysis. The reported normal range of rotation during the CFRT is 44° to each side. A test will be reported as positive when individuals demonstrate a reduction of movement of 10◦ compared to the normal range of motion (<34◦).
Assess the change in Hamstrings flexibility | Before treatment and after 4 weeks treatment
  By Straight leg raising test (SLR) to assess Hamstrings flexibility.The participant will be placed in a supine position, his calcaneus will be held with one hand and the leg will be lifted, and the other hand will be fixed so that the patient's knee is not flexed.

CONTACTS AND LOCATIONS:
Overall Officials: Wadida H Elsayed, Professor, Study Chair — Cairo University; Ghada A Mousa, Ass.prof, Study Director — Cairo University; Hanaa K Atta, Lecturer, Study Director — Cairo University; Nabil H El Agooz, Professor, Study Director — Al-Azhar University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cho SH, Kim SH, Park DJ. The comparison of the immediate effects of application of the suboccipital muscle inhibition and self-myofascial release techniques in the suboccipital region on short hamstring. J Phys Ther Sci. 2015 Jan;27(1):195-7. doi: 10.1589/jpts.27.195. Epub 2015 Jan 9. PMID 25642072